CLINICAL TRIAL: NCT04834024
Title: A Multi-center, Open Label, Phase III Study to Evaluate the Efficacy and Safety of MIL62 Plus Lenalidomide Versus Lenalidomide in Subjects With Follicular Lymphoma Refractory to Rituximab
Brief Title: MIL62 Combined With Lenalidomide Versus Lenalidomide for Patients With Rituximab Refractory Follicular Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIL62-CT301
Record Dates: First submitted 2021-04-05; First posted 2021-04-06 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Follicular Lymphoma and Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Humanized Monoclonal Antibody MIL62, lenalinomide (Experimental)
  Interventions: Drug: Recombinant Humanized Monoclonal Antibody MIL62, lenalinomide
- lenalinomide (Active Comparator)
  Interventions: Drug: lenalinomide

INTERVENTIONS:
Drug: Recombinant Humanized Monoclonal Antibody MIL62, lenalinomide — The patients confirming to the eligibility criteria will receive MIL62 from cycle 1 to cycle 30 and lenalidomide from cycle 1 to cycle 18, unless either rapid disease progression or unacceptable toxicity was observed.
  Arms: Recombinant Humanized Monoclonal Antibody MIL62, lenalinomide
Drug: lenalinomide — The patients confirming to the eligibility criteria will receive lenalidomide for 18 cycles, unless either rapid disease progression or unacceptable toxicity was observed.
  Arms: lenalinomide

SUMMARY:
This phase III trial aims to compare the efficacy and safety of MIL62 combined lenalidomide and lenalidomide alone to treat patient diagnosed with Follicular Lymphoma (FL) and refractory to rituximab. The study randomized patients with a 1:1 ratio to receive either MIL62 plus lenalidomide or lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, >=18 years of age;
2. Patients with either histologically documented CD20-positive FL, WHO grade 1, 2 or 3a
3. Evidence of refractory to rituximab
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
5. At least one bi-dimensionally measurable nodal or tumor lesion defined by CT scan as: greatest transverse diameter > 1.5 cm and a short axis ≥ 10mm
6. Adequate hematologic function
7. Life expectancy >5 years
8. Able and willing to provide written informed consent and to comply with the study protocol

Exclusion Criteria:

1. Evidence of refractory to lenalinomide
2. Central nervous system lymphoma
3. Patients with progressive multifocalleukoencephalopathy (PML)
4. Prior use of any antibody therapy(except for Rituximab ) within 3 months of study start
5. Prior use of any anti-cancer vaccine
6. Prior administration of radiotherapy 42 days prior to study entry
7. Prior administration of chemotherapy 28 days prior to study entry
8. History of prior malignancy within the last 3 years, with the exception of curatively treated basal or squamous cell carcinoma of the skin and low-grade in situ carcinoma of the cervix
9. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
10. Known hypersensitivity to thalidomide or lenalidomide
11. Regular treatment with corticosteroids prior to the start of cycle 1, unless administered for indications other than NHL at a dose equivalent to < 20 mg/day prednisone
12. Any serious active disease or co-morbid medical condition (such as New York Heart Association Class II or IV cardiac disease, severe arrhythmia, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina) or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm or other according to investigator's decision)
13. Infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C(including HBsAg,HBcAb positive with abnormal HBV DAN or HCV RNA )
14. Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (per IRC) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years

SECONDARY OUTCOMES:
Progression-free Survival (per Investigator) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Overall Survival | From date of randomization Until date of death from any cause for up to 5 years
Overall Response Rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Kaplan-Meier Estimate of Duration of Response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Percentage of Participants With Disease Control | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Number of Participants With Treatment Emergent Adverse Events | up to the 1 month the last dose of last subject

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

REFERENCES:
- [Derived] Shi Y, Zhou K, Zhou H, Qin Y, Jing H, Xiang Y, Wang Z, Wang Z, Zang A, Bai O, Li Z, Zhang H, Song Y, Liang J, Wei M. Efficacy and safety of MIL62, a novel glycoengineered type Ⅱ anti-CD20 monoclonal antibody, combined with lenalidomide in patients with relapsed/refractory follicular lymphoma or marginal zone lymphoma: a multicentre, single-arm, phase 1b/2 trial. EClinicalMedicine. 2024 Jun 20;73:102702. doi: 10.1016/j.eclinm.2024.102702. eCollection 2024 Jul. PMID 39007066